CLINICAL TRIAL: NCT05408468
Title: Pilot Evaluation of FAMCOPE-ICU
Brief Title: Pilot Evaluation of FAMCOPE-ICU (Family Coping and Emotion Regulation Tool in the ICU)
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University Hospitals Cleveland Medical Center (Other)
Collaborators: National Center for Advancing Translational Sciences (NCATS) (NIH)
Responsible Party: Principal Investigator, Grant Pignatiello, Instructor and NCATS Clinical Research KL2 Scholar, University Hospitals Cleveland Medical Center
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: STUDY20220055; KL2TR002547 (NIH)
Record Dates: First submitted 2022-06-02; First posted 2022-06-07 (Actual); Results first posted 2025-03-28 (Actual); Last update posted 2025-03-28 (Actual); Status verified 2025-03

CONDITIONS: Emotion Regulation; Coping Skills
Keywords: Critical Care; Informal Caregiving; Surrogate Decision-Making; Self-Regulation
MeSH Terms: conditions — Emotional Regulation; Self-Control

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- FAMCOPE-ICU (Experimental): A digital eHealth emotion regulation and coping intervention.
  Interventions: Behavioral: FAMCOPE-ICU
- Usual Care (No Intervention): The care and support routinely provided to SDMs of critically ill patients.

INTERVENTIONS:
Behavioral: FAMCOPE-ICU — (1) FAMCOPE-ICU is a digital eHealth emotion regulation and coping intervention. FAMCOPE-ICU contains three digital modules representing the three interventional doses. Corresponding with Gross's Extended Process Model of Emotion Regulation, the three respective doses entail assessments, adaptive feedback, and interactive activities pertaining to understanding their affective experiences, learning strategies to regulate emotions and stress, and practicing these skills in a virtual decision-making task. Each dose of the intervention is expected to last 10-15 minutes
  Arms: FAMCOPE-ICU

SUMMARY:
Having a family member or loved one in the ICU can be a very stressful experience. The investigators have created a tablet-based tool (FAMCOPE-ICU) that is designed to help people in this position cope with this experience.

ELIGIBILITY:
Patient Inclusion Criteria:

* 18-89 years old
* Intensive Care Unit (ICU) length of stay (LOS) >= 48 hours
* No anticipated ICU LOS for next 24 hours
* Unable to make healthcare decisions

Family Inclusion Criteria

* Identified by critical care team as legally authorized representative (LAR)
* Able to speak or comprehend English
* >= 18 years old

Patient Exclusion Criteria:

* Less than 18 years or older than 89 years
* ICU LOS < 48 hours
* Anticipated ICU discharge within next 24 hours
* Able to make healthcare decisions

Family Exclusion Criteria

* Not identified by critical care team as the LAR
* Unable to speak or comprehend English
* < 18 years old

Ages: 18 Years to 89 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 49 (Actual)
Dates: Start 2022-08-15 (Actual); Primary Completion 2023-07-27 (Actual); Study Completion 2023-07-27 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Seth A Hoffer, MD, Principal Investigator — University Hospitals Cleveland Medical Center; Grant A Pignatiello, PhD, RN, Principal Investigator — Case Western Reserve University
Locations (1):
- University Hospitals Cleveland Medical Center, Cleveland, Ohio, United States

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: One participant withdrew from study after providing written informed consent, but before baseline data collection.
  The unit of participation was the legally authorized representative for an incapacitated patient.
  Incapacitated patients were not considered enrolled, because our inclusion criteria explicitly required patients to lack capacity to provide consent.
Period: Overall Study
Arm/Group | FAMCOPE-ICU | Usual Care
Started | 29 | 20
Completed | 19 | 17
Not Completed | 10 | 3
Not completed — Lost to Follow-up | 3 | 1
Not completed — Physician Decision | 1 | 0
Not completed — Overwhelmed by clinical situation | 3 | 0
Not completed — Personal illness precluding participation | 1 | 0
Not completed — Withdrawn due to death patient death (unrelated to LAR participation in trial) | 2 | 2

BASELINE CHARACTERISTICS:
Groups:
- FAMCOPE-ICU: A digital eHealth emotion regulation and coping intervention.
  FAMCOPE-ICU: (1) FAMCOPE-ICU is a digital eHealth emotion regulation and coping intervention. FAMCOPE-ICU contains three digital modules representing the three interventional doses. Corresponding with Gross's Extended Process Model of Emotion Regulation, the three respective doses entail assessments, adaptive feedback, and interactive activities pertaining to understanding their affective experiences, learning strategies to regulate emotions and stress, and practicing these skills in a virtual decision-making task. Each dose of the intervention is expected to last 10-15 minutes
  The unit of participation was the legally authorized representative for an incapacitated patient.
- Total: Total of all reporting groups
Arm/Group | FAMCOPE-ICU | Usual Care | Total
Number analyzed (Participants) | 28 | 20 | 48
Age, Continuous [Mean (Standard Deviation); unit: years] | 58.07 (13.84) | 59.20 (12.64) | 58.54 (13.23)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 20 | 16 | 36
  Male | 8 | 4 | 12
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 1 | 0 | 1
  Not Hispanic or Latino | 27 | 20 | 47
  Unknown or Not Reported | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 3 | 4 | 7
  White | 25 | 16 | 41
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0

OUTCOME MEASURES:

1. Primary Outcome: Acceptability of Intervention Measure
Description: Four item self-report survey; item responses range from 1 (completely disagree) to 5 (completely agree)
Time Frame: After dose 1, 5 minutes
Population: Usual care participants did not complete the intervention so no data was collected on them for acceptability of the intervention.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | FAMCOPE-ICU | Usual Care
Number analyzed (Participants) | 24 | 0
units on a scale | 4.36 (0.7) |

2. Primary Outcome: Acceptability of Intervention Measure
Description: Four item self-report survey; item responses range from 1 (completely disagree) to 5 (completely agree)
Time Frame: After dose 2, 5 minutes
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | FAMCOPE-ICU | Usual Care
Number analyzed (Participants) | 24 | 0
units on a scale | 4.37 (0.69) |

3. Primary Outcome: Acceptability of Intervention Measure
Description: Four item self-report survey; item responses range from 1 (completely disagree) to 5 (completely agree)
Time Frame: After dose 3, 5 minutes
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | FAMCOPE-ICU | Usual Care
Number analyzed (Participants) | 19 | 0
units on a scale | 4.27 (1) |

4. Secondary Outcome: Change in Anxiety as Measured by PROMIS Anxiety Short Form
Description: Name: PROMIS Item Bank v1.0-Emotional Distress-Anxiety - Short Form 4a Scoring: The four items' responses (ranging from 1 (Never) to 5 (Always) are summed to form a raw score. The raw scores are converted to a T-Score (mean = 50; Standard deviation = 10) derived from a general population.
  Interpretation: Higher scores indicate a greater severity in anxiety. Scores less than 55 are "within normal limits", 55-60 are "mild", 60-70 are "moderate", and greater than 70 are "severe".
Time Frame: Baseline (enrollment), one week.
Measure: Least Squares Mean (95% Confidence Interval); unit: T score
Arm/Group | FAMCOPE-ICU | Usual Care
Number analyzed (Participants) | 28 | 20
T score
  Baseline | 64.989 [61.521 to 68.457] | 61.30 [57.197 to 64.403]
  One week | 59.394 [55.616 to 63.172] | 57.518 [53.275 to 61.761]
Statistical Analysis 1: Comparison: FAMCOPE-ICU; Test type: Superiority; p = 0.387, Mixed Models Analysis; Mean Difference (Net) = -5.595, Standard Error of Mean 1.731 — Baseline 1.731 One week 1.894
Statistical Analysis 2: Comparison: Usual Care; Test type: Superiority; p = 0.387, Mixed Models Analysis; Mean Difference (Net) = -3.782, Standard Error of Mean 2.048 — Baseline 2.048 One week 2.122

5. Secondary Outcome: Change in Depression as Measured by PROMIS Depression Short Form
Description: Name: PROMIS Item Bank v1.0-Emotional Distress-Depression - Short Form 4a Scoring: The four items' responses (ranging from 1 (Never) to 5 (Always) are summed to form a raw score. The raw scores are converted to a T-Score (mean = 50; Standard deviation = 10) derived from a general population.
  Interpretation: Higher scores indicate greater severity in depression. Scores less than 55 are "within normal limits," 55-60 are "mild," 60-70 are "moderate," and greater than 70 are "severe."
Time Frame: Baseline (enrollment), one week.
Measure: Least Squares Mean (95% Confidence Interval); unit: T Score
Arm/Group | FAMCOPE-ICU | Usual Care
Number analyzed (Participants) | 28 | 20
T Score | 56.896 [53.504 to 60.288] | 53.905 [49.892 to 57.918]
Statistical Analysis 1: Comparison: FAMCOPE-ICU; Test type: Superiority; p = 0.062, Mixed Models Analysis; Mean Difference (Net) = -4.50, Standard Error of Mean 1.693 — Baseline 1.693 One week 1.840
Statistical Analysis 2: Comparison: Usual Care; Test type: Superiority; p = 0.062, Mixed Models Analysis; Mean Difference (Net) = -0.764, Standard Error of Mean 2.003 — Baseline 2.003 One week 2.069

6. Secondary Outcome: Sleep Disturbance as Measured by PROMIS Sleep Disturbance Short Form
Description: Name: PROMIS Item Bank v1.0 - Sleep Disturbance - Short Form 8b Scoring: The eight items' responses (ranging from 1 (Never) to 5 (Always) are summed to form a raw score. The raw scores are converted to a T-Score (mean = 50; Standard deviation = 10) derived from a general population.
  Interpretation: Higher scores indicate greater severity in anxiety. Scores less than 55 are "within normal limits," 55-60 are "mild," 60-70 are "moderate," and greater than 70 are "severe."
Time Frame: Baseline (enrollment)
Measure: Mean (Standard Deviation); unit: T-Score
Arm/Group | FAMCOPE-ICU | Usual Care
Number analyzed (Participants) | 28 | 20
T-Score | 60.63 (8.72) | 55.87 (8.88)

7. Secondary Outcome: Decision Fatigue Scale
Description: Nine item self-report survey; item responses range from 0 (Strongly Disagree) to 3 (Strongly Agree). Item are summed to form a raw score (range 0-27), with higher scores indicated higher decision fatigue.
Time Frame: One week post-enrollment
Measure: Mean (Standard Deviation); unit: Raw score
Arm/Group | FAMCOPE-ICU | Usual Care
Number analyzed (Participants) | 17 | 17
Raw score | 14.47 (10.08) | 11.88 (5.98)
Statistical Analysis 1: Comparison: FAMCOPE-ICU vs Usual Care; Test type: Superiority; p = 0.369, t-test, 2 sided; Median Difference (Final Values) = 2.58, Standard Error of Mean 2.84

8. Secondary Outcome: Decisional Conflict Scale
Description: 10 item self-report survey; item responses are "yes" (0), "unsure" (2), and "no" (4). Items are summed, divided by 10, multiplied by 25. Scores range from 0 (no decisional conflict) to 100 (high decisional conflict)
Time Frame: One week post-enrollment
Measure: Mean (Standard Deviation); unit: Raw score
Arm/Group | FAMCOPE-ICU | Usual Care
Number analyzed (Participants) | 19 | 17
Raw score | 7.89 (13.98) | 5.29 (7.39)
Statistical Analysis 1: Comparison: FAMCOPE-ICU vs Usual Care; Test type: Superiority; p = 0.498, t-test, 2 sided; Median Difference (Final Values) = 2.59, Standard Error of Mean 3.79

9. Secondary Outcome: Satisfaction as Measured by the Family Satisfaction in the Intensive Care Unit Scale - 24R
Description: Four item self-report survey; item responses range from 1 (Very dissatisfied) to 5 (Completely satisfied)
Time Frame: One week post-enrollment
Population: Data not collected, Investigator was concerned about participant burden and ended up not collecting this data. This is a pilot study and this outcome measure was determined to not be worth the participants time.
Arm/Group | FAMCOPE-ICU | Usual Care
Number analyzed (Participants) | 0 | 0

ADVERSE EVENTS:
Time Frame: One week post enrollment
Description: Death was collected as a data point only for the ICU patients related to the LARs. No LARs died from participating in this study. Patient deaths were related to the clinical trajectory and were unrelated to family participation in this study. The unit of participation was the legally authorized representative for an incapacitated patient. Incapacitated patients were not considered enrolled, because our inclusion criteria explicitly required patients to lack capacity to provide consent.
Arm/Group | FAMCOPE-ICU | Usual Care
All-Cause Mortality (participants affected / at risk) | 0/29 | 0/20
Serious Adverse Events (participants affected / at risk) | 0/29 | 0/20
Other Adverse Events (participants affected / at risk) | 0/29 | 0/20

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2022-01-11): https://cdn.clinicaltrials.gov/large-docs/68/NCT05408468/Prot_SAP_000.pdf